# IVROP ReadyforLIFE Program Evaluation Study Protocol

ClinicalTrials.gov ID: NCT05244447

August 29, 2024

# **Descriptive Evaluation Analysis Plan:** "The Evaluation of ReadyforLIFE in Imperial Valley, California"

## A. HMRE grant recipient

HMRE grant recipient: Imperial Valley Regional Occupation Program, El Centro, CA

Project lead: Chantelle Gerardo

Email address: cgerardo@ivrop.org

### **B. Evaluator**

Evaluator's organization: Midwest Evaluation and Research, Emporia, KS

Evaluator lead: McKenna LeClear

Email address: mckenna.leclear@midwestevaluation.com

# Descriptive Evaluation Analysis Plan

# The Evaluation of ReadyforLIFE in Imperial Valley, CA

### A. Description of the intended intervention(s)

The ReadyforLIFE program aims to support the development of healthy, respectful, nonviolent relationships among youth in the Imperial Valley region of California. The primary curriculum includes courses that provide all youth participants with a general overview of healthy partner and family relationships, healthy attitudes and habits about mental health, and money management. Primary workshops are offered predominantly as in-person, in-school sessions that occur during students' regular school hours, though in-person, after school and virtual, evening formats have also been offered to meet the needs of different students. Additionally, participants receive individualized Life Coaching sessions where they can explore career opportunities, get connected to other resources in the community, discuss future interests, and work with their Life Coach to develop an action plan for achieving future goals. A subset of program participants, selected based on their core programming participation and interest on a first-come first-served basis, subject to funding availability, are eligible to receive additional optional program services, described as 2.0 and PLUS services in the outline below. A summary of program services, including dosage and focal population, can be found in Table 1.

- Goal 1 Deliver core curriculum as primary services to all IVROP ReadyforLIFE participants: Participants receive core curriculum to develop healthy attitudes (relationship and financial) and skills to engage in healthy partner and family relationship behaviors, but only after receiving an orientation about the IVROP ReadyforLIFE Program and giving program staff informed consent to participate in study activities. Then, primary ReadyforLIFE curriculum is delivered. Primary curriculum, delivered by an IVROP facilitator, includes 12 hours of Relationship Smarts, 3 hours of Mind Matters, and 1 hour of Money Habitudes, for a total of 16 primary workshop hours, typically delivered sequentially over 4-5 weeks. For in-person, in-school workshops, the number of sessions and length of the workshop series varies depending on classroom schedules. In-school workshops are provided to students whose teachers have agreed to use classroom time to provide the ReadyforLIFE program to their students. ReadyforLIFE is typically offered as a replacement for instructional time in classes that focus on student health and life skills, such as Freshman Seminar, Success 101, or Intro to Health. For in-person and virtual workshops held after school, the delivery schedule is typically as follows:
  - o Relationship Smarts (12 hours total) three 2-hour sessions per week for two weeks
  - Mind Matters (3 hours total) two 1.5-hour sessions held within one week, after the conclusion of Relationship Smarts
  - Money Habitudes (1 hour total) one 1-hour session held either in the same week as Mind Matters or the following week, along with the exit session and makeup workshops as needed

Virtual and in-person afterschool workshops are typically attended by students who do not have teachers who are offering the program as part of the regular school day. Virtual, evening cohorts are typically made up of students who have extracurricular afterschool activities that prevent them from attending in-person, afterschool workshops.

Goal 2 - Deliver support services to all IVROP ReadyforLIFE participants:

Program participants also receive *support services* in the form of individualized life coaching sessions by IVROP facilitators who have been trained in Life Coaching techniques. Life Coaches will offer sessions to build skills to promote independence, decision making, problem solving, and goal setting. Each program participant will be offered at least 3 sessions, to be held virtually or in person. In-person, in-school cohorts are offered Life Coaching services in person, often in a small group setting, and students are able to request 1-on-1 coaching sessions if they prefer. Life Coaching sessions can also be completed on the phone or via Zoom, depending on the needs and preferences of the student.

- Goal 3 Deliver ReadyforLIFE 2.0 Services (Primary + 2.0 services) to a select number of IVROP ReadyforLIFE primary curriculum completers: Program participants, once they complete all primary services (i.e., 16 core curriculum hours), are eligible to receive ReadyforLIFE 2.0 services. Each grant year, 100 students will be offered 2.0 services on a first-come, first-served basis. ReadyforLIFE 2.0 services include the following program activities, with a delivery schedule that varies based on setting:
  - Career Readiness course (6 hours total)
    - In-person, in-school: 1 hour per day for 6 school days
    - Virtual or in-person after school: 2 hours per day for 3 days within 1 week
  - Work-based learning activities with a partner agency (10 hours total) to be completed within 2 weeks outside of school
    - One activity, up to 8 hours (employer-based mentoring OR job shadowing)
      - Employer-based mentoring (either individual or with a small group of participating students) includes discussions about how students can stay on the path toward a particular field (i.e., tips and insights), while job shadowing allows students the opportunity to observe a day in the life of an employee in a particular field
    - One 2-hour activity (employer presentation OR industry tour)
  - At least one additional workshop (time varies based on selection students choose based on their individual interests)
    - Option 1: Developmental Assets course using the Developmental Assets
       Framework curriculum developed by the Search Institute (4 hours total)
      - In-person, in-school: 1 hour per day for 4 school days
      - Virtual or in-person after school: 2 hours per day for 2 days OR
    - Option 2: First5 Parenting workshop using resources developed by First5
       California (8 hours total)
      - In-person, in-school: 1 hour per day for 8 school days
      - Virtual or in-person after school: 2 hours per day for 4 days
    - Participants who are interested in continuing through to ReadyforLIFE PLUS services (Goal 4) must complete both the Developmental Assets and First Five Parenting workshops, as well as the Career Readiness course and work-based learning activities.
- Goal 4 Delivery ReadyforLIFE PLUS Services (Primary, 2.0, and PLUS services) to a select number of ReadyforLIFE Primary and 2.0 curriculum completers: Program participants, once they complete all Primary and 2.0 services (i.e., 16 hours of core curriculum and 28 hours of 2.0 programming), are eligible to receive ReadyforLIFE PLUS services. Each grant year, 35 students who meet these criteria will be offered ReadyforLIFE PLUS services on a first-come, first-served

basis. ReadyforLIFE PLUS services are offered in partnership with employers in the Imperial Valley. Employer partners are identified based on the interests of participating students; IVROP has employer partnerships in agriculture, retail, and health care, among other sectors, and students are able to choose which sectors interest them. ReadyforLIFE PLUS services include the following activities:

- Work-based learning activities with a partner agency (20 hours total, inclusive of 10 hours completed as part of 2.0) to be completed within 4 weeks outside of school
  - Participants will complete all of the work-based learning activities from 2.0 (employer-based mentoring, job shadowing, employer presentation, and industry tour) with a partner agency
- Paid work experience with partner employers (up to 160 hours)
  - During school year maximum of 20 hours per week
  - During summer 40 hours per week for 4 weeks

**Table 1**. Description of intended intervention components, content, dosage and implementation schedule, delivery, and focal populations

| | | Dosage and | | |
|---|---|---|---|---|
| Components | Content | schedule | Delivery | Focal population |
| Relationship skills<br>workshops | Relationships Smarts Plus curriculum: skill- building for youth to have healthy relationships with committed partners | A total of 12 hours, with two-hour sessions occurring three times per week for two weeks (can vary by classroom schedule for inperson, in-school services) | Group classes<br>provided either 1) in-<br>person, in-school, 2)<br>in-person, after<br>school at IVROP<br>facilities, or 3)<br>virtually after school;<br>two trained facilitators<br>lead every session | At-risk youth (defined as attending a high-need high school or meeting other risk criteria such as membership in a low-income or single parent household) ages 14-18 and enrolled in 9-12 <sup>th</sup> grades |
| Mental health<br>workshops | Mind Matters curriculum: skill- building that helps youth resolve ACEs to manage emotions and improve their state of mind | A total of three hours,<br>with two 1.5-hour<br>sessions held within<br>one week | Group classes<br>provided either 1) in-<br>person, in-school, 2)<br>in-person, after<br>school at IVROP<br>facilities, or 3)<br>virtually after school;<br>two trained facilitators<br>lead every session | At-risk youth (defined as attending a high-need high school or meeting other risk criteria such as membership in a low-income or single parent household) ages 14-18 and enrolled in 9-12 <sup>th</sup> grades |
| Economic stability<br>workshops | Money Habitudes curriculum: skill-building that uses personality types to develop better money attitudes and habits | A total of one hour,<br>with one 1-hour<br>session held in the<br>same week as Mind<br>Matters or the<br>following week | Group classes<br>provided either 1) in-<br>person, in-school, 2)<br>in-person, after<br>school at IVROP<br>facilities, or 3)<br>virtually after school;<br>two trained facilitators<br>lead every session | At-risk youth (defined as attending a high-need high school or meeting other risk criteria such as membership in a low-income or single parent household) ages 14-18 and |

| Components | Content | Dosage and schedule | Delivery | Focal population |
|---|---|---|---|---|
| | | | | enrolled in 9-12 <sup>th</sup><br>grades |
| Life coaching<br>sessions | Individualized sessions to promote independence, decision making, problem solving, and goal setting | At least three 1-hour sessions | Individual sessions provided by IVROP-trained Life Coaches either virtually or in person | At-risk youth (defined as attending a high-need high school or meeting other risk criteria such as membership in a low-income or single parent household) ages 14-18 and enrolled in 9-12 <sup>th</sup> grades |
| ReadyforLIFE 2.0 (optional, secondary for up to 100 students per grant year) | Career readiness<br>course; work-based<br>learning activities;<br>parenting or<br>developmental assets<br>course provided by<br>IVROP facilitators | A total of 20-28 hours<br>(depending on<br>selections; course<br>schedule can vary by<br>classroom schedule<br>for in-person, in-<br>school services) | Group classes provided either 1) in- person, in-school, 2) in-person, after school at IVROP facilities, or 3) virtually after school; group work-based learning activities with partner employers or IVROP's Strong Workforce agency | At-risk youth (defined as attending a high-need high school or meeting other risk criteria such as membership in a low-income or single parent household) ages 14-18 and enrolled in 9-12 <sup>th</sup> grades who complete all ReadyforLIFE primary services |
| ReadyforLIFE Plus<br>(optional, secondary<br>for up to 35 students<br>per grant year) | Work-based learning<br>activities; paid work<br>experience | Up to 180 hours total, with a maximum of 20 hours per week of paid work experience during the school year and a maximum of 40 hours per week of paid work experience during the summer | Individual/group work-based learning activities and individual paid work with partner employers | At-risk youth (defined as attending a high-need high school or meeting other risk criteria such as membership in a low-income or single parent household) ages 14-18 and enrolled in 9-12 <sup>th</sup> grades who complete all ReadyforLIFE primary and 2.0 services |

**Table 2**. Staff education and training (initial and ongoing)

| Component | Education and initial training | Ongoing training |
|---|---|---|
| Relationship skills<br>workshops | Facilitators: 1 male and 4 females All facilitators hold a bachelor's degree and received 5 days (17.5 hours) of initial training. | Receive yearly refresher trainings during seasonal breaks to include, school's thanksgiving and summer breaks, and attend semiannual content webinars that cover curriculum enhancements offered by the Dibble Institute. |

| Component | Education and initial training | Ongoing training |
|---|---|---|
| Mental health<br>workshops | Facilitators: 1 male and 4 females All facilitators hold a bachelor's degree and received 5 days (17.5 hours) of initial training. | Receive yearly refresher trainings during seasonal breaks to include, school's thanksgiving and summer breaks, and attend semiannual content webinars. |
| Economic stability workshops | Facilitators: 1 male and 4 females All facilitators hold a bachelor's degree and received 2 days (5 hours) of initial training. | Receive yearly refresher trainings during seasonal breaks to include, school's thanksgiving and summer breaks, and attend semiannual content webinars. |
| Life coaching<br>sessions | Facilitators: 1 male and 4 females All facilitators hold a bachelor's degree and received 30 contact hours of Life Coach training for certification, in addition to completing 20 practicum hours. | Receive yearly refresher trainings during seasonal breaks to include, school's thanksgiving and summer breaks, and attend semiannual content webinars. |
| Career readiness<br>workshops | Facilitators: 1 male and 4 females All facilitators hold a bachelor's degree and received 3 days (6 hours) of initial training. | Receive yearly refresher trainings during seasonal breaks to include, school's thanksgiving and summer breaks, and attend semiannual content webinars. |
| Developmental<br>Assets workshops<br>(for 2.0 participants<br>only) | Facilitators: 1 male and 4 females All facilitators hold a bachelor's degree and received an initial curriculum training | Receive yearly refresher trainings from<br>Search Institute during seasonal breaks to<br>include schools' Thanksgiving and summer<br>breaks |
| First5 Parenting<br>workshops (for 2.0<br>participants only) | Facilitators: 1 male and 4 females All facilitators hold a bachelor's degree and received an initial training with First5 California | IVROP staff who received the initial training from First5 conduct train-the-trainer refreshers among staff |

#### **B.** Outcomes study

This section describes the research questions, evaluation enrollment process, data collection procedures, outcome measures, and analytic approach for the outcomes study.

#### 1. Research questions

RQ1: What is the level of healthy relationship attitude scores immediately following ReadyforLIFE primary services, as compared to baseline scores?

RQ2: What is the level of healthy relationship behavior scores one year after enrollment into ReadyforLIFE primary services, as compared to baseline scores?

RQ3: What is the level of healthy financial attitude scores immediately following ReadyforLIFE primary services, as compared to baseline scores?

RQ4: What is the level of healthy financial behavior scores one year after enrollment into ReadyforLIFE primary services, as compared to baseline scores?

#### 2. Outcomes evaluation enrollment

The original study and data collection plan were initially approved by Solutions IRB on 3/30/2021 and have been annually reviewed and approved three times on 3/15/2022, 3/4/2023, and 3/11/2024.

Additionally, revisions to the study and/or data collection plan were submitted to the IRB as amendments and were approved on 4/6/2022 and 2/22/2023.

All program participants whose parents have given consent are eligible to participate in the evaluation study. Participants for the ReadyforLIFE program, and thus the study, are recruited primarily from partnerships with schools and particular teachers in the Imperial Valley region who have agreed to offer ReadyforLIFE programming as part of their classroom instructional time. IVROP staff give presentations to school administrators and directly to students to foster interest in the program. Monthly presentations directly to students in classrooms generate an interest list that IVROP uses to fill after school and summer workshops. Program service locations participating in the local evaluation since the start of the program have included:

- Brawley Union High School
- Central Union High School
- Calipatria High School
- Southwest High School
- Holbrook High School
- Desert Valley High School
- Renaissance High School
- Phoenix Rising High School
- After-school services provided at IVROP facilities
- Virtual services provided via Zoom

The projected enrollment into the study is 1680 participants, and the desired sample size, with a target follow-up survey response rate of 70%, is 1176 participants.

To be eligible for the program, and thus the study, participants must meet the following criteria: 1) at-risk youth (e.g., former foster care system involved, runaways, homeless, low income, migrant, at risk for dropping out of school, expecting or parenting teens, or attending a Title 1 or alternative high school), 2) ages 14-18, 3) parents have given consent for youth to participate, and 4) youth have given assent to participate in the study. All students offered services in a classroom setting meet the first criterion, as services are offered in Title 1 or alternative high schools. Enrolling students are also asked to identify if they meet other risk criteria (e.g., low-income household, single parent household, etc.). Eligibility for virtual and after school workshops is determined by the IVROP program manager using responses on the enrollment packet paperwork.

Parental consent for enrollment into the evaluation is collected as part of the program enrollment process. A consent form explaining study activities and potential risks and benefits is provided to parents as part of the enrollment packet with information on who to contact with questions. Parents who wish to

deny consent for their youth to be part of the study will sign and return the form to program staff. Youth assent for enrollment into the evaluation happens during program orientation, prior to the start of the first primary workshop. The study activities and potential risks and benefits are explained to the youth, who have an opportunity to opt out of the local evaluation. Consent records are kept on MER's secure Dropbox server.

Enrollment into the study began on June 15, 2021 and is expected to continue until March 31, 2024, after which point study enrollment will end to allow for collection of the one-year follow-up survey before final analyses and report writing begin in 2025.

#### 3. Data sources and data collection

The main data source for this study is surveys of intervention participants. Participants are surveyed at three different time points throughout the study. Two surveys (one nFORM and one local evaluation [OLLE] survey) are collected from participants at each of the first two waves of data collection. Wave 1 (nFORM entrance survey and OLLE pre-survey) of data collection happens during the program orientation session before the first primary workshop session, with make-ups administered as needed until three primary workshops have been received. Wave 2 (nFORM exit survey and OLLE post-survey) of data collection happens at or immediately after the final workshop session, with make-ups administered as needed for up to two weeks after primary workshops end. Wave 3 of data collection (the OLLE follow-up survey) happens one year after program enrollment.

Waves 1 and 2 of surveys are administered online using students' school computers, program tablets, or students' personal devices in the case of virtual cohorts. Paper surveys can be offered if necessary due to technological difficulties or facility restrictions. The link to complete the follow-up survey at Wave 3 is sent to participants via email, text message, and postcard/letter using a QR code. Participants can also complete the survey over the phone with evaluation team staff if they prefer.

Wave 1 of data collection began in June 2021 and will conclude at the end of March 2024. Wave 2 of data collection began in July 2021 and is expected to conclude in April 2024. Wave 3 of data collection began in June 2022 and is expected to conclude in March-April 2025.

The analyses for this study will use data from different survey waves, depending on the outcome. Short-term attitudinal changes will be assessed by comparing outcomes between Waves 1 and 2 (program entry to exit), and longer-term behavioral changes will be assessed by comparing outcomes between Waves 1 and 3 (program entry to follow-up).

A copy of the local evaluation survey codebook will be sent as a separate appendix to this plan.

**Table 3**. Sources of data to address the research questions

| Data source | Timing of data collection | Mode of data collection | Start and end date of data collection |
|---|---|---|---|
| Intervention<br>participants<br>(nFORM entrance<br>survey and OLLE<br>pre-survey) | At the orientation session before<br>the first primary workshop | In-person online survey or remote online survey | June 2021-March 2024 |

| Data source | Timing of data collection | Mode of data collection | Start and end date of data collection |
|---|---|---|---|
| Intervention<br>participants<br>(nFORM exit and<br>OLLE post-survey) | At or immediately after the final primary workshop session with make-ups offered as needed | In-person online survey or remote online survey | August 2021-May 2024 |
| Intervention participants (OLLE follow-up survey) | One year after program enrollment | Remote online survey sent via text, email, or QR code; phone survey | June 2022-March 2025 |

#### 4. Outcome measures

The attitudinal research questions for this study will be answered by comparing post-survey responses collected at the end of primary workshop services to baseline survey responses collected before primary workshops begin. The behavioral research questions for this study will be answered by comparing follow-up survey responses collected one year after program enrollment to baseline survey responses collected before primary workshops begin. The one-year follow-up survey will be administered to all program participants who consent to be in the study and complete at least one baseline survey (nFORM or OLLE), regardless of program completion status or workshop delivery format. Because the post-surveys (nFORM exit and OLLE post-survey) are collected during or shortly after the final primary workshop, it is likely that only those complete the program will complete the post-surveys; however, all study participants who have consented and completed at least one baseline survey are eligible to take the post-surveys.

For each outcome construct (healthy relationship attitudes, healthy relationship behaviors, healthy financial attitudes, and healthy financial behaviors), we have identified the relevant survey measures that are theoretically aligned with that construct. When analysis begins, we will generate a correlation matrix between items in a given construct to ensure that theoretically related items are also empirically related in our data set. Survey items will be reverse-coded as needed before checking for correlation strength. Items that are not strongly correlated with other items in a construct will be removed as necessary. Factor analysis will be used to ensure that all construct items hang together, using an alpha of 0.7 or higher as the acceptable threshold. If a constructed scale does not achieve an alpha of 0.7 or higher, even after removing items that are not well correlated, the outcome measure will be dropped from the analysis.

We will then create a composite measure for each construct by taking an average of the scores on each non-missing item in the construct. For these composite measures, we intend to use 20% as a threshold for allowable missing items; this plan is contingent on the final distribution of missing data in our data set. Participants who are missing more than 20% of items for a given construct will be assigned a missing value for that composite outcome measure. We will not be imputing truly missing values for outcomes. To create the construct score for each participant, the average of the relevant survey items will be divided by the number of non-missing values in the construct.

**Table 4**. Outcomes used to answer the research questions

| Research question | Outcome name | Description of the outcome measure | Source of the measure | Timing of measure |
|---|---|---|---|---|
| RQ1 | Healthy<br>relationship<br>attitudes | The outcome measure is a scale (value range 1-4) calculated as the average of nine survey items related to healthy relationship beliefs | nFORM entrance<br>survey (A1.a-i);<br>nFORM exit survey | Wave 1 (before<br>primary workshops<br>begin) and Wave 2<br>(at the final primary<br>workshop) |
| RQ1 | Healthy<br>relationship<br>attitudes | The outcome measure is a scale (value range 1-5) calculated as the average of three survey items related to expectations that youth have for their future relationship circumstances | nFORM entrance<br>survey (A2.a-c);<br>nFORM exit survey | Wave 1 (before<br>primary workshops<br>begin) and Wave 2<br>(at the final primary<br>workshop) |
| RQ2 | Healthy<br>relationship<br>behaviors | The outcome measure is a scale (value range 1-4) calculated as the average of five survey items related to reported self-assessed skill with communication and conflict resolution | nFORM entrance<br>survey (C1b.a-e);<br>OLLE follow-up<br>survey | Wave 1 (before<br>primary workshops<br>begin) and Wave 3<br>(one year after<br>program enrollment) |
| RQ2 | Healthy<br>relationship<br>behaviors | The outcome measure is a scale (value range 1-5) calculated as the average of six survey items related to the frequency of engaging in unhealthy conflict resolution behaviors | nFORM entrance<br>survey (C3.a-f);<br>OLLE follow-up<br>survey | Wave 1 (before primary workshops begin) and Wave 3 (one year after program enrollment) |
| RQ3 | Healthy financial attitudes | The outcome measure is a scale (value range 1-5) calculated as the average of seven survey items related to level of agreement with key financial attitudes | OLLE pre-survey<br>(Q14.a-g); OLLE<br>post-survey | Wave 1 (before primary workshops begin) and Wave 2 (at the final primary workshop) |
| RQ4 | Healthy financial<br>behaviors | The outcome measure is a scale (value range 1-5) calculated as the average of four survey items related to level of agreement with good money management habits | OLLE pre-survey<br>(Q21.a-d); OLLE<br>follow-up survey | Wave 1 (before primary workshops begin) and Wave 3 (one year after program enrollment) |